CLINICAL TRIAL: NCT06300203
Title: The Efficacy and Safety of Humanized Antibody Targeting the Interleukin-4 Receptor Alpha Subunit (IL-4Rα) in Patients With Uncontrolled Seasonal Allergic Rhinitis Under Standard Treatment： A Randomized, Double-Blind, Placebo-controlled IIT Study
Brief Title: Study of CM310 in Patients With Uncontrolled Seasonal Allergic Rhinitis
Acronym: MEGREZ
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310_IIS_SAR07
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interleukin-4 receptor responders (Experimental): Interleukin-4 receptor was injected subcutaneously.
  Interventions: Biological: Interleukin-4 receptor responders
- Placebo (Placebo Comparator): Placebo was injected subcutaneously.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Interleukin-4 receptor responders — Interleukin-4 receptor was injected subcutaneously.
  Arms: Interleukin-4 receptor responders
Other: Placebo — Placebo was injected subcutaneously.
  Arms: Placebo

SUMMARY:
Allergic rhinitis (AR) is a non-infectious chronic inflammatory disease of the nasal mucosa mainly mediated by immunoglobulin E after exposure to allergens in atopic individuals. The typical symptoms of AR are paroxysmal sneezing, watery rhinorrhea, itching, and nasal congestion, which may be accompanied by ocular symptoms, including eye itching, tearing, redness, and burning sensation, which are more common in patients with hay fever allergies. Bronchial asthma is associated with bronchial asthma in 40% of patients with AR, suggesting a comorbid feature of allergic disease.

DETAILED DESCRIPTION:
AR is a common clinical chronic nasal disease, affecting 10% to 20% of the world's population, and has become a global health problem. AR not only seriously affects the quality of life of patients, resulting in patient fatigue, impaired learning, attention, and decision-making ability, but also causes a heavy social burden.

AR has a variety of classification methods. According to the type of allergen, it can be divided into seasonal (SAR, common allergens are seasonal allergens such as pollen) and perennial (PAR, common allergens are indoor allergens such as dust mites or occupational allergies), which is a classification method often used in clinical studies. According to the course of the disease, it can be divided into intermittent (symptom onset < 4 days/week, or < 4 consecutive weeks) and persistent (symptom onset ≥ 4 days/week, and ≥ 4 consecutive weeks). According to the severity of the disease, it can be divided into minor AR (mild symptoms, with no significant impact on quality of life) and moderate-severe AR (more severe or severe symptoms, with significant impact on quality of life). The results of the cooperative survey showed that persistent moderate-to-severe disease was the most common in the overall population, accounting for 52.2%, indicating that the treatment and control of AR has become an urgent problem to be solved.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Have any condition that are not suitable for participating in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Average change from baseline in daily retrospective total nasal symptom score (rTNSS) at week 2. | up to Week 2
  Average change from baseline in daily retrospective total nasal symptom score (rTNSS) during treatment period. The Total Nasal Symptom Score (TNSS) is the sum of the four symptom scores of runny nose, nasal congestion, nasal itching, and sneezing, with each symptom scoring from 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Study Chair — Beijing Tong-Ren hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No